CLINICAL TRIAL: NCT06576596
Title: Apnoeic Oxygenation During Pediatric Tracheal Intubation: a Study Protocol for a Single-center, Cluster Randomized Clinical Trial (ApOx-Pedi-Trial)
Brief Title: Apnoeic Oxygenation During Pediatric Tracheal Intubation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. med. Davut Deniz Uzun, Resident Departement of Anesthesiology, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ApOxHeidelberg
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia; Airway Complication of Anesthesia; Anesthesia; Adverse Effect
Keywords: Airway Management; Pediatric Anesthesia; Apnoeic Oxygenation; Apneic Oxygenation; Oxygen; Tracheal Intubation

STUDY DESIGN:
Intervention Model Description: prospective, monocentric, single-blinded clinical trial. Intervention group: receive apnoeic oxygenation via the nose Control group: Does not receive apnoeic oxygenation (standard care)
Who Masked: Participant, Outcomes Assessor
Masking Description: The parents and the child are completely blinded to the study (Child is under anaesthesia, parents are not in the operating theatre). The study is also analysed by a blinded employee of Heidelberg University Hospital, Germany.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard induction of anaesthesia in the child. (No Intervention): Control group: in this group, standard induction of anaesthesia is performed without the use of apnoeic oxygenation.
- Experimental group: standard induction is supplemented by apnoeic oxygenation. (Experimental): In the experimental group, apnoeic oxygenation is used in addition to standard anaesthesia induction.
  Interventions: Other: apnoeic Oxygenation

INTERVENTIONS:
Other: apnoeic Oxygenation — One approach to preventing adverse respiratory events due to hypoxaemia during paediatric anaesthesia is the use of apnoeic oxygenation. The principle is to deliver oxygen to the airways of anaesthetised patients via a conventional nasal cannula. As less carbon dioxide is produced than oxygen is consumed during apnoea, the supply of oxygen to the upper airways leads to an 'inward diffusion' of oxygen, which may prolongs the time until desaturation and hypoxaemia occur.
  Arms: Experimental group: standard induction is supplemented by apnoeic oxygenation.

SUMMARY:
The goal of this randomized, controlled, single-blinded clinical trial is to evaluate the effectiveness of apnoeic Oxygenation in pediatric anesthesia. The main question it aims to answer are:

primary outcome measure: The primary outcome will be the lowest SpO₂ value recorded during the apnoeic period.

secondary outcome measure:

* Differences in intubation first-pass-success (key secondary objective)
* Temporal differences to achieve successful intubation
* Differences in time to oxygen desaturation
* Differences in heart rate and mean arterial blood pressure decrease
* Differences in the incidence of anesthesia-related adverse events

The study participants are randomized two age dependents groups. Either in the control group without the use of apnoeic oxygenation or in the intervention group with the use of apnoeic oxygenation.

The study population will be divided into two independent cohorts, each consisting of 100 patients. The first cohort, designated as "infants" will include all patients aged up to 24 months, while the second cohort, termed "children" will comprise patients aged older than 24 months and up to six years.

Within each cohort, patients will be randomized into an intervention group and a control group, with 50 patients assigned to each. This randomization will ensure that, for both the Infant and Children Groups, half of the participants (n=50) will receive the intervention, while the other half (n=50) will serve as controls.

Statistical analysis of primary and secondary endpoints will be conducted independently for each cohort. This stratified approach will allow for targeted evaluation of age-specific effects of the intervention, as well as comparison between intervention and control outcomes within each age-defined cohort.

DETAILED DESCRIPTION:
The incidence of intraoperative hypoxaemia in children is high and age-dependent. An incidence of over 10 % is reported in8- to 16-year-old children and over50 % in newborns. Severe respiratory critical events occur in paediatric anaesthesia with an incidence of 3.1 %. After the onset of apnoea, hypoxaemia develops more rapidly in children than in adults, which is due to increased oxygen consumption, a lower functional residual capacity and an increased closing capacity. These events can lead to permanent neurological damage or death. One approach to preventing adverse respiratory events due to hypoxaemia during paediatric anaesthesia is the use of apnoeic oxygenation. The principle is to supply oxygen to the airways of anaesthetised patients via a conventional nasal cannula. As less carbon dioxide is produced than oxygen is consumed during apnoea, the supply of oxygen to the upper airways leads to an 'inward diffusion' of oxygen, which prolongs the time until desaturation and hypoxaemia occur. This also extends the 'safe apnoea time' and the anaesthetist has more time to secure the airway. As the incidence and severity of arterial oxygen desaturation is higher in critically ill children compared to healthy children, this vulnerable group in particular could benefit from apnoeic oxygenation. Apnoeic oxygenation is increasingly becoming a standard technique in paediatric anaesthesia, with applications ranging from induction of anaesthesia in the operating theatre and standard airway management to the management of difficult airways. In its current guidelines, the European Society of Anaesthesiology and Intensive Care recommends the use of apnoeic oxygenation in the airway management of newborns and infants. The main aim of this study is to evaluate the effectiveness of apnoeic oxygenation in terms of time to desaturation and hypoxaemia, as well as the impact of apnoeic oxygenation on intubation success in anaesthetised children.

ELIGIBILITY:
Inclusion Criteria:

* children 0-6 years
* ASA status I-III
* Elective surgery/intervention under general anaesthesia

Exclusion Criteria:

* refusal to participate in the study by the patients or their legal guardians
* ASA classification IV = patients with life-threatening disease
* Existing oxygen therapy prior to surgery
* Surgery/intervention in the ENT area with contraindication for oxygen goggles
* Injuries/trauma in the ENT and mouth/nose area
* Anatomical anomalies/malformations in the ENT and mouth/nose area
* Chronical hypoxemia (e.g. patients with cyanotic heart diseases)
* language barrier (parent/guardian)
* emergency interventions
* refusal by the attending physician
* lack of presence of the pediatric anesthesiology consultant
* Situational inability to perform apnoeic oxygenation or inability to obtain baseline NIRS values at room air within 60 seconds from the first attempt due to agitation of the patient

Ages: 0 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the lowest SpO₂ value recorded during the apnoeic period. | The time frame refers only to the induction of anaesthesia and subsequent airway management.
  The main aim of anaesthesia is to avoid a drop in saturation during induction of anaesthesia. This time until the drop in oxygen saturation is described as the so-called 'safe apnoea time'.

SECONDARY OUTCOMES:
Differences in intubation first-pass-success (key secondary outcome) | The time frame refers only to the induction of anaesthesia and subsequent airway management.
  Differences in the 'first-pass-succes' of intubation between the two groups are highlighted here.
Temporal differences to achieve successful intubation | The time frame refers only to the induction of anaesthesia and subsequent airway management.
  Comparison of the time differences for a successful intubation.
Differences in time to oxygen desaturation | The time frame refers only to the induction of anaesthesia and subsequent airway management.
  Comparison of the time differences to desaturation.
Differences in heart rate and mean arterial blood pressure decrease | The time frame refers only to the induction of anaesthesia and subsequent airway management.
  Comparison of the differences in heart rate and arterial blood pressure between the groups.
Differences in the incidence of anesthesia-related adverse events | The time frame refers only to the induction of anaesthesia and subsequent airway management.
  Comparison of the differences of anesthesia-related adverse events between the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty Heidelberg, Department of Anesthesiology, Heidelberg University,, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
This aspect is still being clarified with the competent authority and will be announced in due course.

REFERENCES:
- [Derived] Uzun DD, Zimmermann BP, Knoeller S, Kirchner M, Mohr S, Weigand MA, Zivkovic AR, Schmitt FCF. Apnoeic oxygenation during paediatric tracheal intubation: a study protocol for a single-centre, cluster randomised clinical trial (ApOx-Pedi-Trial). BMJ Open. 2025 May 2;15(5):e096842. doi: 10.1136/bmjopen-2024-096842. PMID 40316345